CLINICAL TRIAL: NCT00577369
Title: A Pilot Study to Measure Blood Levels of Desflurane in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Anesthesiology Associates, Ltd. (Other)
Responsible Party: Kha Tran, MD, The Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-12-5096
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Desflurane Levels
Keywords: arterial line; end-expiratory desflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): The subject's participation will take place over one surgical procedure. It will begin with the first blood collection and end with either the second blood draw or the end of the procedure.
  Interventions: Other: Desflurane Levels

INTERVENTIONS:
Other: Desflurane Levels — The subject's participation will take place over one surgical procedure. It will begin with the first blood collection and end with either the second blood draw or the end of the procedure.

SUMMARY:
In this feasibility study we will collect blood from indwelling arterial catheters in up to 20 patients undergoing non-emergent surgery with desflurane anesthesia at Children's Hospital of Philadelphia. Desflurane levels will be determined by high pressure liquid chromatography (HPLC).

Our eventual goal is to quantify fetal levels of desflurane in umbilical cord blood during fetal surgery. We propose a pilot study to assess the ability of our assay to measure desflurane in human blood.

DETAILED DESCRIPTION:
Fetal surgery is an evolving field. Some previously fatal diseases can be surgically corrected before birth. Animal models of the procedures have been carefully translated to humans, but less is known about anesthetic techniques. In children, inadequate anesthesia results in greater stress responses as shown by cardiovascular, neuro-endocrine, and metabolic changes. These stress responses have been associated with poorer outcomes. One of the major goals of anesthesia for these procedures is to attenuate this stress response. Fetuses get intramuscular opioids before their incision, and the mother is given high doses of volatile anesthetic (desflurane) with the assumption that whatever amount of desflurane crosses the placenta adequately anesthetizes the fetus. No studies have quantified the fetal levels of desflurane.

High pressure liquid chromatography (HPLC) has been used to measure levels of volatile anesthetic in various tissues. Measurement of desflurane has been challenging because of its higher boiling point (23.5 °C at one atmosphere pressure) when compared to older volatile anesthetics such as sevoflurane (boiling point 58.6 °C) and isoflurane (boiling point 48.5 °C). With techniques in cold rooms and using ice for sample transport, investigators have successfully measured desflurane levels in blood and brain tissue of mice.

Our eventual goal is to quantify fetal levels of desflurane in umbilical cord blood during fetal surgery, but we first propose a pilot study to assess and refine the ability of our assay to measure desflurane in human blood.

ELIGIBILITY:
Inclusion Criteria:

1. Children between 1 and 18 years old
2. Weight >10 kg
3. Scheduled for elective surgery
4. Patient will have an arterial catheter placed as routine care for the surgery
5. Informed consent (and assent if applicable)

Exclusion Criteria:

1. Desflurane not used as part of anesthetic
2. Preoperative hemoglobin less than 9 mg/dl
3. Any investigational drug use within 30 days prior to enrollment
4. Pregnant or lactating females

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will simply be the successful measurement of desflurane in human blood. | During one operation.

SECONDARY OUTCOMES:
Secondary endpoints will include obtaining similar levels of desflurane across several patients who are have similar levels of end expiratory desflurane. | During one operation.

CONTACTS AND LOCATIONS:
Overall Officials: Kha Tran, MD, Principal Investigator — Children's Anesthesiology Associates, Ltd.
Locations (1):
- The Children's Hospital Of Philadelphia, Philadelphia, Pennsylvania, United States